CLINICAL TRIAL: NCT06945432
Title: Comparing 68Ga-CTR-FAPI and 18F-FDG PET/ CT in Cancer Detection
Status: Completed | Type: Observational
Sponsor: Lanzhou University Second Hospital (Other)
Responsible Party: Principal Investigator, Yuxi Zhang, Dr., Lanzhou University Second Hospital
Other Study IDs: YZhang
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-02

CONDITIONS: Tumors; PET / CT; FDG PET/CT; FAPI
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to compare the diagnostic efficacy of 68Ga-CTR-FAPI PET/CT and 18F-FDG PET/CT in various malignant tumors

DETAILED DESCRIPTION:
This study recruited malignant tumor patients diagnosed by histopathology and imaging at the Nuclear Medicine Department of Lanzhou University Second Hospital from July 2024 to March 2025. The enrolled patients underwent 68Ga-CTR-FAPI PET/CT and 18F-FDG PET/CT scans within one week.

ELIGIBILITY:
Inclusion Criteria:

(a) Age ≥ 18 years old; (b) Suspected or newly diagnosed malignant tumors, evaluating the therapeutic effect of the tumor, or discovering recurrence/metastasis; (c) Obtain approval from oncologists and agree to undergo 18F-FDG and 68Ga-CTR-FAPI PET/CT scans within one week.

Exclusion Criteria:

(a) Pregnancy or lactation period; (b) Claustrophobia. (c) Serious health problems: such as severe heart, liver and kidney dysfunction, diseases that affect the metabolism or clearance of imaging agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Malignant tumor patients diagnosed by histopathology and imaging
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Lesion uptake | 1 day
  Standardized uptake value (SUV)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Lanzhou University, Lanzhou, Gansu, China